CLINICAL TRIAL: NCT05898451
Title: Effect of Refnot on Immunity in Cancer Patients
Acronym: R-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Refnot-Pharm Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2
Record Dates: First submitted 2023-05-18; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Solid Tumor
Keywords: solid tumors; Refnot
MeSH Terms: interventions — Drug Therapy; Dacarbazine; Lomustine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Independent use of Refnot (Experimental): Refnot is administered at a dose of 400,000 IU subcutaneously 3 times a week for 4 weeks. 4 weeks constitute 1 course of treatment with Refnot. In the absence of progression of the disease - an additional 4 weeks.
  Interventions: Drug: Tumor necrosis factor-thymosin alfa 1 recombinant (TNF-T)
- The use of Refnot in combination with chemotherapy (Experimental): Refnot is administered at a dose of 400,000 IU subcutaneously 3 times a week for 4 weeks. 4 weeks constitute 1 course of treatment with Refnot. In the absence of progression of the disease - an additional 4 weeks. Chemotherapy may be used after 4-8 weeks of Refnot use.
  Interventions: Drug: Tumor necrosis factor-thymosin alfa 1 recombinant (TNF-T) and chemotherapy

INTERVENTIONS:
Drug: Tumor necrosis factor-thymosin alfa 1 recombinant (TNF-T) — has a direct antitumor effect in vitro and in vivo on various tumor cell lines
  Other Names: Refnot; Tumor necrosis factor-thymosin alfa 1 recombinant
  Arms: Independent use of Refnot
Drug: Tumor necrosis factor-thymosin alfa 1 recombinant (TNF-T) and chemotherapy — Refnot has a direct antitumor effect in vitro and in vivo on various tumor cell lines, chemotherapy has a cytostatic and cytotoxic effect.
  Other Names: and Dacarbazine, Lomustine, Cisplatin
  Arms: The use of Refnot in combination with chemotherapy

SUMMARY:
The study was planned to include disseminated patients with various solid tumors (melanoma, soft tissue sarcoma, breast cancer, colon cancer, etc.). The study drug was administered subcutaneously at a dose of 400,000 IU once a day, 3 times a week (every other day), for 4 weeks. In the absence of disease progression - an additional 4 weeks.

DETAILED DESCRIPTION:
The study was planned to include 50 disseminated patients with various solid tumors. The patients were divided into 2 groups: 1 - Refnot, monotherapy, 2 - Refnot together with chemotherapy.

Refnot is administered at a dose of 400,000 IU subcutaneously 3 times a week for 4 weeks. 4 weeks constitute 1 course of treatment with Refnot. Immediately before use, 1 ml of water for injection is added to 4 vials (100,000 IU each) or to a vial containing 400,000 IU. After dilution, the drug is injected subcutaneously into the outer surface of the shoulder or thigh. Injection sites should alternate. In the absence of progression of the disease - an additional 4 weeks. Chemotherapy may be used after 4-8 weeks of Refnot use.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have exhausted standard methods of treatment.
* Morphological (histological or cytological) confirmation of the diagnosis.
* Age no more than 75 years.
* General condition 0-2 (WHO).
* Estimated life expectancy of at least 3 months.
* Consent to treatment under this protocol.
* The number of granulocytes is more than 2000/mm, platelets are more than 150000/mm.
* The level of creatinine should not exceed 1.5 norms, liver enzymes (ALT, AST and alkaline phosphatase) should not exceed 3 norms.
* For common disease, patients should receive standard treatment earlier.

Exclusion Criteria:

* Severe manifestations of cardiovascular diseases in the past and at present (myocardial infarction, hypertension, stroke, phlebothrombosis, coronary insufficiency requiring drug control, etc.).
* Peptic ulcer of the stomach, duodenal ulcer (in the acute phase), uncorrected diabetes mellitus.
* Mental illness preventing understanding of the treatment plan.
* Pregnancy.
* Metastases of a malignant tumor in the brain (according to clinical data).
* Chronic use of corticosteroids or immunosuppressants.
* Various neurological diseases that prevent this treatment.
* Known allergic reactions and/or other significant allergic conditions.
* Any immunotherapy within the last 6 weeks prior to enrollment in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-06-04 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in the level of CD3+-cells | 4 weeks
  An increase in the level of CD3+-cells relative to the initial
Change in the level of CD4+-cells | 2 weeks
  An increase in the level of CD4+-cells relative to the initial
Change in the level of CD4+-cells | 4 weeks
  An increase in the level of CD4+-cells relative to the initial
Change in the level of CD8+-cells | 2 weeks
  An increase in the level of T-lymphocytes relative to the initial one in those patients in whom it was reduced
Change in the level of CD8+-cells | 2 weeks
  A decrease in the level of T-lymphocytes relative to the initial one in those patients in whom it was elevated
Change in the ratio of CD4+/CD8+ | 2 weeks
  Increase in the ratio of lymphocytes / lymphocytes relative to the initial
Change in the ratio of CD4+/CD8+ | 4 weeks
  Increase in the ratio of lymphocytes / lymphocytes relative to the initial
Change in NK-cell activity | 4 weeks
  Increased activity of NK cells in patients with an initially reduced rate
Change in NK-cell activity | 2 weeks
  Percentage increase in NK cell activity in patients with initially normal values
Change in NK-cell activity | 4 weeks
  Percentage increase in NK cell activity in patients with initially normal values

CONTACTS AND LOCATIONS:
Overall Officials: Anatolij D Namgaladze, Master, Study Director — Refnot-Pharm Ltd